CLINICAL TRIAL: NCT02941354
Title: A Multicentre, Open-label Trial Evaluating the Pharmacokinetics of NovoEight® (Turoctocog Alfa) in Relation to BMI in Subjects With Haemophilia A
Brief Title: Evaluating the Pharmacokinetics of NovoEight® (Turoctocog Alfa) in Relation to BMI in Subjects With Haemophilia A
Acronym: guardian ™9
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-4239; 2015-004379-56 (EudraCT Number); U1111-1175-1191 (Other: WHO)
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Turoctocog alfa (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Each subject will receive a single dose of turoctocog alfa as an intravenous (i.v.) bolus injection of 50 IU/kg.

SUMMARY:
This trial is conducted globally. The aim of this trial is evaluating the pharmacokinetics (the exposure of the trial drug in the body) of NovoEight® (turoctocog alfa) in relation to BMI (body mass index) in subjects with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male, age at least 18 years at the time of signing informed consent
* History of more than 150 exposure days to any factor VIII products
* Subjects with the diagnosis of congenital haemophilia A with factor VIII activity below 1%, based on medical records

Exclusion Criteria:

* Known history of factor VIII inhibitors
* Inhibitors to factor VIII (above or equal to 0.6 BU (Bethesda units)) at screening measured by the Nijmegen modified Bethesda method
* Known congenital or acquired coagulation disorders other than haemophilia A
* Previous participation in pharmacokinetic sessions with turoctocog alfa in another trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Plasma FVIII activity at 30 minutes(C30min) | At 30 minutes post-dose
  Based on samples taken at pre-dose (-1hour), 15minutes, 30minutes, 1hour, 3hours, 6hours, 9hours, 24hours, 28hours, 48hours, 72hours post-dose

SECONDARY OUTCOMES:
Area under the FVIII activity-time curve | From 0 up to 72 hours after administration
Incremental recovery FVIII at 30 minutes (IR30min) | At 30 minutes post-dose
  Based on samples taken at pre-dose (-1hour), 15minutes, 30minutes, 1hour, 3hours, 6hours, 9hours, 24hours, 28hours, 48hours, 72hours post-dose
Terminal half-life (t½) of FVIII | From 0 up to 72 hours after administration
Clearance (CL) of FVIII | From 0 up to 72 hours after administration
Apparent volume of distribution at steady state (Vss) of FVIII | From 0 up to 72 hours after administration

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Germany (2):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Hanover
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Spain (4):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Vigo
- Taiwan (2):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com